CLINICAL TRIAL: NCT06262022
Title: The Effect of Cold Application on Pain Level, Edema and Drainage Amount in Patients With Total Knee Arthroplasty: A Randomized Controlled Study
Brief Title: The Effect of Cold Application on Pain Level, Edema and Drainage Amount
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma GÖK, lecturer, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KaramanogluMehmetbeyUFGok
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Cold Therapy; Pain, Postoperative
Keywords: cold therapy; pain; patient; knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: This study was planned as a prospective, parallel, two-arm (1:1) randomized controlled trial (RCT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): A cold ice pack will be applied to the patient's knee for 20 minutes every hour for three days, starting after total knee arthroplasty.
  Interventions: Other: cold therapy
- control arm (No Intervention): Only unit-specific routine treatment and care interventions will be applied to the patients in the control arm by the team in the unit, and no intervention will be applied by the researcher.

INTERVENTIONS:
Other: cold therapy — A cold ice pack will be applied to the patient's knee for 20 minutes every hour for three days, starting after total knee arthroplasty.
  Arms: experimental arm

SUMMARY:
In this study, we aimed to investigate the effect of cold application applied for 20 minutes every hour for 8 hours on the first day, second and third days after total hip arthroplasty with gel pads, on the pain level, edema and drainage amount of total hip arthroplasty patients. The main question[s]it aims to answer are:

* Is there a difference between the pain levels of patients in the control and cold application arms?
* Is there a difference between the knee edema of patients in the control and cold application arms?
* Is there a difference between the amount of drainage of patients in the control and cold application arms? This study was planned as a prospective, parallel, two-arm (1:1) randomized controlled trial (RCT).

DETAILED DESCRIPTION:
* When the patient arrives at the service after TKA, cold application will begin with gel pads at 0 ºC and continue for eight hours. After TKA, cold application will continue for 20 minutes every hour between 08.00-16.00 on the 1st and 2nd day.
* After TKA, pain intensity will be evaluated and at the 6th, 24th and 48th hours.
* Knee circumference measurements for knee edema will be made before TKA and at the 24th and 48th hours after TKA.
* After being taken to bed after TKA, the amount of drainage will be measured at the 1st, 6th and 24th hours.
* In the first 24 hours and 24-48 hours after TKA. Analgesic consumption between hours will be recorded.
* Knee temperature will be measured before and after each cold application.
* Knee temperature will be measured before and after each cold application. Measurements of the control group will be made at the specified times in the cold application group. Cold application will not be applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above,
* Able to communicate verbally and in writing,
* Turkish speaking,
* TKA applied for the first time,
* Unilateral total knee arthroplasty applied,
* Spinal anesthesia applied,
* Having a hemovac drainage catheter,
* Without peripheral vascular disease,

Exclusion Criteria:

* Revision total knee arthroplasty applied,
* Bilateraltotal knee arthroplasty applied,
* Those who use alcohol and substances,
* TKA was performed for a reason other than knee osteoarthritis,
* General anesthesia applied,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
pain level | After total knee arthroplasty, pain intensity will be evaluated at the 6th, 24th and 48th hours.
  Pain level of patients will be measured after total knee arthroplasty ( Visual Analogue Scale (VAS) is a 10 cm ruler with "no pain" written on one end and "the worst possible pain" written on the other end. Patients mark the levels on the ruler according to their pain levels. 1-3 points on the scale are rated as mild, 4-6 points as moderate and 7-10 points as severe pain.)

SECONDARY OUTCOMES:
edema | Knee circumference measurements for knee edema will be made before total knee arthroplasty and at the 24th and 48th hours after total knee arthroplasty.
  The knee circumference of patients will be measured before total knee arthroplasty and will be measured again at 24 and 48 hours after surgery.
amount of drainage | After being taken to bed after total knee arthroplasty, the amount of drainage will be measured at the 1st, 6th and 24th hours.
  The amount coming from the drain after total knee arthroplasty will be measured

OTHER OUTCOMES:
Analgesic consumption | The first 24 hours and 24-48 hours after total knee arthroplasty. Analgesic consumption between hours will be recorded.
  The type and amount of analgesics used by patients after total knee arthroplasty will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoğlu Mehmet bey Üniversitesi, Merkez, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No